CLINICAL TRIAL: NCT03549611
Title: Randomized Comparison of Two Pre-induction Analgesia Regimens: Multimodal vs Acetaminophen in the Reduction of Post-operative Pain Following Ureteroscopy With Lithotripsy for Kidney Stones Evaluated With Text Messaging
Brief Title: Pre-induction Analgesia: Multimodel Regimen vs Aceteminophen for Post Ureteroscopy Pain
Acronym: MMPITR
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: elected not to proceed with the study
Sponsor: Kevin J Flynn MD (Other)
Responsible Party: Sponsor-Investigator, Kevin J Flynn MD, Urology Resident, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201805826
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Kidney Calculi; Pain, Postoperative
Keywords: ureteroscopy; opioids; narcotics; text messaging; real time data acquisition; ecologic momentary assessments; pre-emptive analgesia; gabapentin; meloxicam; tamsulosin; kidney stones; lithotripsy; nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Pain, Postoperative; Nephrolithiasis | interventions — Gabapentin; Oxycodone; Acetaminophen; Celecoxib

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient will not be made aware which treatment regimen they are receiving and neither will the attending urologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Multimodel Drug Regimen (Experimental): The patients randomized to this arm will receive the following multimodal oral drug regimen administered shortly before induction of general anesthesia
  1. Tylenol, 975mg (3 tabs)
  2. 800mg Gabapentin
  3. 400mg Celecoxib
  4. 10mg Oxycodone
  Interventions: Drug: Multimodal Oral Drug Regimen
- Acetaminophen Only (Active Comparator): The patients randomized to this arm will receive oral acetaminophen only administered shortly before induction of general anesthesia
  1. Tylenol, 975mg (3 tabs)
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Multimodal Oral Drug Regimen — Regimen of 4 pharmacologic agents that provides analgesia by acting on 4 different physiologic pain pathways
  Other Names: Gabapentin 800mg; Oxycodone 10mg; Acetaminophen 975mg; Celecoxib 400mg
  Arms: Multimodel Drug Regimen
Drug: Acetaminophen — Acetaminophen 975mg
  Other Names: Tylenol
  Arms: Acetaminophen Only

SUMMARY:
Adult patients with kidney stones undergoing surgical intervention with ureteroscopy with laser lithotripsy will be randomized to receive one of two different regimens of oral medications administered prior to induction of general anesthesia. Postoperatively, patients will receive automated daily text messages to assess pain and opioid consumption and subsequently determine which which treatment regimen is superior.

DETAILED DESCRIPTION:
Adult patients undergoing ureteroscopy for kidney stones will be screened and those who meet initial study criteria (adult, English speaking, non-pregnant, non-intellectually disabled patients), will be sent an information letter outlining the study. Interested patients, who possess a phone capable of text messaging will be consented to enroll in the study and randomized to one of two preoperative analgesic treatment arms (see below) that will be administered in the preoperative area prior to induction of general anesthesia.

Multimodal Analgesia Arm

1. Acetaminophen 975mg
2. Gabapentin 800mg
3. Oxycodone 10mg
4. Celecoxib 400mg

Acetaminophen Only Analgesia Arm

a. Acetaminophen 975mg

Consenting patients will fill out a baseline demographics questionnaire as well as provide baseline levels of pain and opioid consumption prior to surgery. They will also be enrolled to receive automated postoperative pain assessments and opioid consumption inquiries via text message. The patients will be blinded to the treatment they are receiving. The research team will not be blinded. The patient will then proceed with their planned ureteroscopy. The patient will then undergo their planned ureteroscopy with lithotripsy for kidney stone disease; the study does not change any parameters about the surgery itself. The general anesthesia regimen will be standardized to one particular standard of care method so as to minimize the potential effect of confounders.

All patients (patients in both preoperative analgesia treatment regimen arms) will be monitored in the post-anesthesia recovery unit for pain, blood pressure, sedation level monitored by the Ramsey Sedation Scale. Once they have recovered appropriately and met standard discharge criteria they will be discharged with the following analgesic regimen

1. Tylenol 650 every 6 hours x 7 day
2. Oxybutynin 5mg three times daily as needed for x 7 days
3. Flomax 0.4mg daily x 7 days
4. Oxycodone, 5mg as needed 15 pills
5. Celecoxib daily for 7 days

Patients will receive a pain assessment via text message the evening of postoperative day 0, and then twice a day for 14 days. Patients will also receive an opioid consumption inquiry once a day for 14 days. On postoperative day 15 patients will be asked if they were happy with their postoperative pain control.

During the study period the research team will access the patients electronic medical record to review and record the following information

* Current medications
* height, weight, age, gender, marital status, city, state of residence
* Co-morbid medical conditions
* insurance
* stone parameters: size (mmm), location, laterality, number of stones,
* Operative factors: instruments used, operative time, operative complications
* post-operative course: emergency department visits, unexpected phone calls, unexpected clinic visits, other 30-day complications

ELIGIBILITY:
Inclusion Criteria:

* Adult Patient (greater than 18 years old)
* Possesses or has access to cell phone with text message capability
* Undergoing ureteroscopy with lithotripsy for a ureteral or kidney stones

Exclusion Criteria:

* Does not possess or have access to a cell phone with text message capability
* Non-English speaking
* Incarcerated individuals
* undergoing planned secondary procedure
* pregnancy
* intellectual disability
* History of, anaphylactic, rash, or other hypersensitivity reaction to any of the study agents
* Patients with history of CABG, myocardial infarction, endovascular cardiac stent, gastrointestinal bleed, or gastric ulcer disease will not receive Celecoxib. They may still participate in the study otherwise, it will be documented that they did not receive an NSAID component.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative day 0 Pain | 4-6 hours after conclusion of surgery
  The magnitude of pain (0-10) that the patient experiences in the evening after their surgery concludes

SECONDARY OUTCOMES:
Time to pain resolution | Approximately the first 72-96 hours
  The amount of time (days) that it takes for patients to report a pain level of less than 4 (0-10 scale)
Opioid Consumption | 14 days following surgery
  The number of total opioid pills a patient consumes following surgery
Time to complete pain resolution | 14 days
  The amount of time (days) that it takes for patients to report a pain level of 0 (0-10 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Tracy, MD, Principal Investigator — University of Iowa Department of Urology

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

REFERENCES:
- [Background] Ahn ST, Kim JH, Park JY, Moon du G, Bae JH. Acute postoperative pain after ureteroscopic removal of stone: incidence and risk factors. Korean J Urol. 2012 Jan;53(1):34-9. doi: 10.4111/kju.2012.53.1.34. Epub 2012 Jan 25. PMID 22323972
- [Background] Penprase B, Brunetto E, Dahmani E, Forthoffer JJ, Kapoor S. The efficacy of preemptive analgesia for postoperative pain control: a systematic review of the literature. AORN J. 2015 Jan;101(1):94-105.e8. doi: 10.1016/j.aorn.2014.01.030. PMID 25537330
- [Background] Scales CD Jr, Smith AC, Hanley JM, Saigal CS; Urologic Diseases in America Project. Prevalence of kidney stones in the United States. Eur Urol. 2012 Jul;62(1):160-5. doi: 10.1016/j.eururo.2012.03.052. Epub 2012 Mar 31. PMID 22498635
- [Background] Oberlin DT, Flum AS, Bachrach L, Matulewicz RS, Flury SC. Contemporary surgical trends in the management of upper tract calculi. J Urol. 2015 Mar;193(3):880-4. doi: 10.1016/j.juro.2014.09.006. Epub 2014 Sep 16. PMID 25219700
- [Background] Barnes KT, Bing MT, Tracy CR. Do ureteric stent extraction strings affect stent-related quality of life or complications after ureteroscopy for urolithiasis: a prospective randomised control trial. BJU Int. 2014 Apr;113(4):605-9. doi: 10.1111/bju.12541. PMID 24765679
- [Background] Hirschtritt ME, Delucchi KL, Olfson M. Outpatient, combined use of opioid and benzodiazepine medications in the United States, 1993-2014. Prev Med Rep. 2017 Dec 21;9:49-54. doi: 10.1016/j.pmedr.2017.12.010. eCollection 2018 Mar. PMID 29340270